CLINICAL TRIAL: NCT05776992
Title: Effect of Different Virtual Reality Exercise in Nonspecific Individuals With Low Back Pain
Brief Title: Effect of Various Virtual Reality Exercise Individuals With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, physiotherapist PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Virtual Reality Application
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prior to and following the eight-week application, evaluation was conducted
Who Masked: Investigator
Masking Description: Treatment and assessment in the study was performed by different physiotherapists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balance games (Experimental): virtual reality games
  Interventions: Device: Xbox virtual reality games
- balance training (Active Comparator): Biodex balance training
  Interventions: Device: Biodex balance training

INTERVENTIONS:
Device: Xbox virtual reality games — X-box balance evaluation was implemented in a completely dark and isolated room specially prepared for this treatment and evaluation
  Arms: balance games
Device: Biodex balance training — the Biodex Balance System SD has been designed to meet the needs of everyone looking to improve balance, increase agility, develop muscle tone and treat a wide variety of pathologies.
  Arms: balance training

SUMMARY:
Posture is defined as the best position formed by the segments that make up the body in a harmonious arrangement with each other. Muscle strength, which is one of the primary factors in providing a static or dynamic posture, is achieved thanks to the antigravity muscles that keep the body upright against gravity. Proper posture is ensured by a good body balance.

DETAILED DESCRIPTION:
Advances in technology can influence healthcare providers to create alternative and new treatment options. SG/LV applications have also gained momentum in the field of rehabilitation. Studies have shown that 12-week programs, especially in diseases affecting the balance and vestibular system, can achieve more effective results than standard physiotherapy programs in both upper and lower extremity functions, balance, walking parameters, fall risk and cognitive parameters. The use of popular video game-based exercises, such as XBOX, or "exergaming," has evolved to become therapeutic tools for rehabilitation. Accessible as technology evolves into more and more, equipment like biodex could be an alternative way to assess and train balance

ELIGIBILITY:
Inclusion Criteria:

* 18-60 with nonspecific chronic low back pain

Exclusion criteria from the study:

* Cognitive impairment
* Disc herniation
* Neurological deficit
* Respiratory problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-07-02 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | 6 weeks
  The Visual Analogue Scale (VAS) was used to evaluate the severity of pain, and the patients were asked to mark the level of pain they felt before and after the treatment. The VAS is a 10-centimeter straight line, the number 0 (zero) at one end indicates no pain, and the number 10 (ten) at the other end represents unbearable pain. The points marked by the patients were measured with the help of a ruler starting from the 0 point and recorded as numerical values.
Y Balance Test | 6 weeks
  Y balance test, a large Y tape is drawn on the flat surface such that the angle between the front and back directions is 135 degrees, and the angle between the two back sides is 90 degrees. The person is asked to place their feet exactly in the center. It is explained that while balancing on one foot, she/he should reach anterior (front), posterolateral (posterior external), and posteromedial (posterior internal) directions with the other foot, and keep her/his weight on a stable foot. Three attempts are made before starting the test
Oswestry Low Back Pain Disability Questionnaire | 6 weeks
  It is a questionnaire that aims to evaluate the disability levels and quality of life faced by patients due to low back pain. It includes 1 item related to pain and 9 items related to activities of daily living (personal care, lifting, walking, sitting, standing, sleep, sexual life, social life and travel). Each item is measured on a 6-point rank scale between 0 and 5 points according to the scenarios it contains. At the end of the survey, the scores are summed and the percentage value is calculated for the total score. High score indicates poor functional level.
Algometer | 6 weeks
  The Algometer used (JTECH Medical-Algometer Commander-USA, Electronic Algometer) is a digital algometer with an LCD display, which can be used as a wrist unit or desktop system, and where measurements can be made in kilograms or Newtons.
Body Awareness Questionnaire | 6 weeks
  In 13 statements, some situations in which people feel about themselves are listed. After reading each statement, they are asked to write the number in the space to the left of the statement, evaluating from 1 to 7 the degree to which the statement is true for them.
Flamingo Static Balance Evaluation Test: | 6 weeks
  Flamingo balance test (FBT) is a test used for balance measurements in the Eurofit test battery.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Dayanir IO, Birinci T, Kaya Mutlu E, Akcetin MA, Akdemir AO. Comparison of Three Manual Therapy Techniques as Trigger Point Therapy for Chronic Nonspecific Low Back Pain: A Randomized Controlled Pilot Trial. J Altern Complement Med. 2020 Apr;26(4):291-299. doi: 10.1089/acm.2019.0435. Epub 2020 Feb 5. PMID 32023423